CLINICAL TRIAL: NCT01288833
Title: Real Time Colorectal Polyp Diagnosis in Colorectal Cancer Screening Using Close Focus High Definition Narrow Band Imaging Colonoscopy Compared to Conventional Histopathology Diagnosis - the VALID (Veterans Affairs Lesion Interpretation and Diagnosis) Colonoscopy Study
Brief Title: Clinical Study of Real Time Colorectal Polyp Diagnosis During Colonoscopy - the VALID Colonoscopy Study
Acronym: VALID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Roy Soetikno, Co-Principal Investigator, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: VALID PA19624
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Neoplasm; Colonic Polyps
Keywords: Colonoscopy; Diagnostic Imaging; Colorectal Neoplasm; Primary Prevention; Cost and Cost Analysis; Endoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Close focus HD NBI Colonoscopy System (Experimental): Use of close focus to make optical diagnosis
  Interventions: Device: Close focus HD NBI Colonoscopy System
- Current HD NBI Colonoscopy System (No Intervention): Use of standard focus for optical diagnosis

INTERVENTIONS:
Device: Close focus HD NBI Colonoscopy System — Technically improved colonoscope with close focus high definition narrow band imaging. Optical specifications include a 2mm near field focal depth.
  Arms: Close focus HD NBI Colonoscopy System

SUMMARY:
The investigators hypothesize that high definition colonoscopy with close focus narrow band imaging features has a high diagnostic accuracy for colorectal polyp histology, and can replace formal pathologic assessment in cases of high diagnostic confidence.

DETAILED DESCRIPTION:
A recent single arm prospective cohort study suggested that high definition colonoscopy with narrow band imaging is an acceptable strategy to diagnose polyp histology and determine future surveillance intervals. Endoscopic proficiency in macroscopic features to differentiate polyp histology can be attained in a relatively short time period. A new high definition colonoscope with close focus narrow band imaging features may further improve diagnostic accuracy for polyp differentiation, and can replace formal pathologic assessment in cases of high diagnostic confidence.

Primary Aim: Compare the diagnostic accuracy of high definition narrow band imaging colonoscopy with and without close focus features for the macroscopic differentiation of neoplastic and non-neoplastic colorectal lesions using histopathologic diagnosis as the reference standard.

Secondary Aims: Compare diagnostic characteristics of the colonoscopes, measure concordance of high confidence and accuracy, compare accuracy of predicted versus actual surveillance interval recommendations, perform a cost-effective analysis of endoscopic versus pathologic diagnoses, and measure complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients referred for routine colonoscopy

Exclusion Criteria:

* Known inflammatory bowel disease
* Personal or family history of polyposis or non-polyposis syndrome
* Presentation for emergency endoscopy
* Inability to remove polyp due to coagulopathy or thrombocytopenia
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2011-03; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Kaltenbach, MD MS, Principal Investigator — Veterans Affairs Palo Alto; Roy Soetikno, MD MS, Principal Investigator — Veterans Affairs Palo Alto
Locations (2):
- United States (2):
  - Veterans Affairs Palo Alto, Palo Alto, California
  - Veterans Affairs Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaltenbach T, Sano Y, Friedland S, Soetikno R; American Gastroenterological Association. American Gastroenterological Association (AGA) Institute technology assessment on image-enhanced endoscopy. Gastroenterology. 2008 Jan;134(1):327-40. doi: 10.1053/j.gastro.2007.10.062. Epub 2007 Oct 30. PMID 18061178
- [Background] Muto M, Katada C, Sano Y, Yoshida S. Narrow band imaging: a new diagnostic approach to visualize angiogenesis in superficial neoplasia. Clin Gastroenterol Hepatol. 2005 Jul;3(7 Suppl 1):S16-20. doi: 10.1016/s1542-3565(05)00262-4. PMID 16012987
- [Background] Rex DK. Narrow-band imaging without optical magnification for histologic analysis of colorectal polyps. Gastroenterology. 2009 Apr;136(4):1174-81. doi: 10.1053/j.gastro.2008.12.009. Epub 2008 Dec 10. PMID 19187781
- [Background] Raghavendra M, Hewett DG, Rex DK. Differentiating adenomas from hyperplastic colorectal polyps: narrow-band imaging can be learned in 20 minutes. Gastrointest Endosc. 2010 Sep;72(3):572-6. doi: 10.1016/j.gie.2010.03.1124. Epub 2010 Jun 19. PMID 20561618
- [Background] Rastogi A, Keighley J, Singh V, Callahan P, Bansal A, Wani S, Sharma P. High accuracy of narrow band imaging without magnification for the real-time characterization of polyp histology and its comparison with high-definition white light colonoscopy: a prospective study. Am J Gastroenterol. 2009 Oct;104(10):2422-30. doi: 10.1038/ajg.2009.403. Epub 2009 Jul 7. PMID 19584829
- [Background] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250
- [Background] Rex DK, Fennerty MB, Sharma P, Kaltenbach T, Soetikno R. Bringing new endoscopic imaging technology into everyday practice: what is the role of professional GI societies? Polyp imaging as a template for moving endoscopic innovation forward to answer key clinical questions. Gastrointest Endosc. 2010 Jan;71(1):142-6. doi: 10.1016/j.gie.2009.09.011. Epub 2009 Nov 17. No abstract available. PMID 19922926
- [Derived] von Renteln D, Kaltenbach T, Rastogi A, Anderson JC, Rosch T, Soetikno R, Pohl H. Simplifying Resect and Discard Strategies for Real-Time Assessment of Diminutive Colorectal Polyps. Clin Gastroenterol Hepatol. 2018 May;16(5):706-714. doi: 10.1016/j.cgh.2017.11.036. Epub 2017 Nov 23. PMID 29174789
- [Derived] Kaltenbach T, Rastogi A, Rouse RV, McQuaid KR, Sato T, Bansal A, Kosek JC, Soetikno R. Real-time optical diagnosis for diminutive colorectal polyps using narrow-band imaging: the VALID randomised clinical trial. Gut. 2015 Oct;64(10):1569-77. doi: 10.1136/gutjnl-2014-307742. Epub 2014 Nov 11. PMID 25387891
- [Derived] McGill SK, Soetikno R, Rastogi A, Rouse RV, Sato T, Bansal A, McQuaid K, Kaltenbach T. Endoscopists can sustain high performance for the optical diagnosis of colorectal polyps following standardized and continued training. Endoscopy. 2015 Mar;47(3):200-6. doi: 10.1055/s-0034-1378096. Epub 2014 Sep 29. PMID 25264764

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Close Focus HD NBI Colonoscopy System | Current HD NBI Colonoscopy System
Started | 277 | 281
Completed | 277 | 281
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Close Focus HD NBI Colonoscopy System | Current HD NBI Colonoscopy System | Total
Number analyzed (Participants) | 277 | 281 | 558
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (7.7) | 62.4 (8.7) | 62.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 261 | 269 | 530
Indication [Count of Participants; unit: Participants]
  Screening | 104 | 106 | 210
  Surveillance | 121 | 123 | 244
  Symptoms | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Rate of Accurate High Confidence Polyp Histology Predictions by the Endoscopist in the Two Groups.
Description: Measure of the percentage of accurate high confidence predictions by the endoscopist in the differentiation of neoplastic from non-neoplastic colorectal lesions, using the high definition NBI colonoscopy with and without close focus features. High confidence was assigned if the polyp had one or more features of Type 2 (neoplasia) or Type 1 (nonneoplasia) in the NICE classification and no features associated with the other histology Note: one patient may have multiple polyps.
Time Frame: At the time of procedure
Population: We analyzed all diminutive sized polyps to assess the number of polyps that endoscopists were able to make an accurate high confidence optical diagnosis. High confidence was assigned if the polyp had one or more features of Type 2 (neoplasia) or Type 1 (non-neoplasia) in the NICE classification and no features associated with the other histology.
Measure: Number (95% Confidence Interval); unit: Percent of accurate HC predictions
Units Other Than Participants: Polyps analyzed
Arm/Group | Close Focus HD NBI Colonoscopy System | Current HD NBI Colonoscopy System
Number analyzed (Participants) | 277 | 281
Number analyzed (Polyps analyzed) | 530 | 445
Percent of accurate HC predictions | 75.3 [71.3 to 78.9] | 63.1 [58.5 to 67.6]

2. Secondary Outcome: Cost
Description: Measure the cost of colonoscopy with macroscopic histopathologic diagnosis of colorectal lesions compared to colonoscopy with conventional microscopic histopathologic diagnosis, on the lesions that were managed based on an accurate endoscopic diagnosis.
  A reduction in pathology specimens may improve the efficiency of the procedure and has direct pathology cost savings (as well as indirect savings, which were not measured).
Time Frame: At the time of procedure
Measure: Number; unit: Specimen bottles that could be omitted
Arm/Group | Close Focus HD NBI Colonoscopy System | Current HD NBI Colonoscopy System
Number analyzed (Participants) | 277 | 281
Specimen bottles that could be omitted | 241 | 0

3. Secondary Outcome: Diagnostic Characteristics
Description: Compare the diagnostic characteristics (sensitivity, specificity, positive predictive value and negative predictive value) using the high definition narrow band imaging colonoscopy with and without close focus features.
  Accuracy: number of endoscopic predictions of adenomatous polyps histologically confirmed to be adenomatous/number of predicted hyperplastic polyps confirmed to be hyperplastic out of all polyps Sensitivity: number of endoscopic predictions (optical diagnosis) of adenomatous (neoplastic) polyps out of all histologically confirmed polyps Specificity: number of endoscopic predictions of hyperplastic (non-neoplastic) polyps out of all histologically confirmed polyps PPV: number of histologically confirmed adenomatous polyps out of all endoscopic predictions of adenomatous polyps NPV: number of histologically confirmed hyperplastic polyps out of all endoscopic predictions of hyperplastic (non-neoplastic) polyps Note: a patient may have multiple polyps
Time Frame: At time of procedure
Population: 975 total polyps were found with high confidence predictions made on 774 of them.We assessed diagnostic performance of the high confidence predictions. High confidence was assigned if the polyp had one or more features of Type 2 (neoplasia) or Type 1 (nonneoplasia) in the NICE classification and no features associated with the other histology.
Measure: Number (95% Confidence Interval); unit: percentage of high confidence prediction
Units Other Than Participants: Polyps analyzed
Arm/Group | Close Focus HD NBI Colonoscopy System | Current HD NBI Colonoscopy System
Number analyzed (Participants) | 277 | 281
Number analyzed (Polyps analyzed) | 451 | 323
percentage of high confidence prediction
  Accuracy | 88.5 [85.2 to 91.3] | 87.0 [82.8 to 90.5]
  Sensitivity | 98.2 [95.5 to 99.3] | 95.2 [90.8 to 97.6]
  Specificity | 73.9 [66.7 to 80] | 75.7 [67.5 to 82.5]
  PPV | 85.0 [80.5 to 88.8] | 84.4 [78.7 to 89.0]
  NPV | 96.4 [91.8 to 98.8] | 92.0 [85.3 to 96.3]

4. Secondary Outcome: Accuracy of Predicted Versus Actual Surveillance Intervals
Description: Compared the accuracy of predicted versus actual surveillance colonoscopy interval recommendations by determining number of patients with correct surveillance interval recommendation.
Time Frame: At the time of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Close Focus HD NBI Colonoscopy System | Current HD NBI Colonoscopy System
Number analyzed (Participants) | 277 | 281
Participants
  Predicted (optical diagnosis) | 259 | 259
  Actual (histopathological diagnosis) | 277 | 281

5. Secondary Outcome: Learning Curve
Description: Examine the impact of a learning curve (i.e. NPV of high confidence at each of endoscopist's first 50% of exams versus last 50% exams to endoscopically predict polyp histology). NPV is defined as "number of histologically confirmed hyperplastic polyps out of all endoscopic predictions of hyperplastic (non-neoplastic) polyps.
Time Frame: At time of procedure.
Population: 975 total polyps were found and we were able to make high confidence predictions on 774 of them.
Measure: Number (95% Confidence Interval); unit: percentage of high confidence prediction
Units Other Than Participants: Diminutive polyps
Arm/Group | Close Focus HD NBI Colonoscopy System | Current HD NBI Colonoscopy System
Number analyzed (Participants) | 277 | 281
Number analyzed (Diminutive polyps) | 530 | 445
percentage of high confidence prediction
  First half | 94.9 [87.5 to 98.6] | 88.0 [75.7 to 95.5]
  Second half | 96.7 [88.5 to 99.6] | 95.8 [88.3 to 99.1]

6. Post Hoc Outcome: Surveillance Colonoscopy Advanced Pathology Findings
Description: Compare the advanced pathology and colon cancer incidence at surveillance colonoscopy of the groups who underwent high definition narrow band imaging colonoscopy with and without close focus features, and more specifically who underwent macroscopic versus microscopic polyp management. This applies if we bring the patient back after 5 years, we have not collected the data yet.
Time Frame: 5 to 10 years after colonoscopy
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Close Focus HD NBI Colonoscopy System | Current HD NBI Colonoscopy System
Serious Adverse Events (participants affected / at risk) | 0/277 | 0/281
Other Adverse Events (participants affected / at risk) | 0/277 | 0/281

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No